CLINICAL TRIAL: NCT00395265
Title: Association of Thrombophilia and Inflammation With Post-Thrombotic Syndrome
Brief Title: Evaluating the Relationship Between Blood Clotting Disorders, Inflammation, and Obesity in Individuals With Venous Disorders and Post-Thrombotic Syndrome
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Mary Cushman, Professor of Medicine and Pathology, University of Vermont
Other Study IDs: 1342; R01HL083926 (NIH); HL083926
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Venous Thrombosis; Venous Insufficiency
Keywords: Deep Vein Thrombosis; Chronic Venous Insufficiency; Post Thrombotic Syndrome; Blood Coagulation; Inflammation
MeSH Terms: conditions — Venous Thrombosis; Venous Insufficiency; Postthrombotic Syndrome; Thrombosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Venous thrombosis is the development of a blood clot in a vein. Post-thrombotic syndrome (PTS) is a painful condition that can develop following a venous thrombosis in one of the deep veins of the leg. While PTS is mainly thought to occur because of damage to the vein, other factors may be responsible for the development of this condition. This study will analyze genetic and biologic samples from participants of a previous study to examine other possible causes of venous diseases and PTS.

DETAILED DESCRIPTION:
The long-term effects of venous thrombosis, known collectively as PTS, include persistent swelling, pain, cramps, and numbness in the leg. These symptoms result from impaired return of blood through the veins of the lower leg to the heart. PTS is believed to occur as a result of direct damage to the valves and walls of the vein. There may be specific factors that make certain individuals more prone to PTS. Individuals who are obese, have a genetic predisposition to blood clotting disorders, or have high levels of inflammation biomarkers may have an increased risk of developing venous diseases. The purpose of this study is to investigate the possible link between these factors and the occurrence of chronic venous disease and PTS. The study's findings will be useful in developing new prevention and treatment strategies.

This study will examine previously collected data from participants in the San Diego Population Study, a study that gathered information on the prevalence of chronic venous disease in a multi-ethnic group of individuals. There will be no study visits specifically for this study. Researchers will examine stored genetic and biologic samples of 370 control participants and 370 participants with chronic venous disease. Specifically, levels of inflammation biomarkers, levels of obesity-related biomarkers, and genetic predispositions for blood clotting disorders will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the San Diego Population Study

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will examine previously collected data from participants in the San Diego Population Study.
Sampling Method: Non-Probability Sample
Enrollment: 2211 (Actual)
Dates: Start 2006-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cushman, MD, MSc, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

REFERENCES:
- [Background] Criqui MH, Jamosmos M, Fronek A, Denenberg JO, Langer RD, Bergan J, Golomb BA. Chronic venous disease in an ethnically diverse population: the San Diego Population Study. Am J Epidemiol. 2003 Sep 1;158(5):448-56. doi: 10.1093/aje/kwg166. PMID 12936900